CLINICAL TRIAL: NCT00552253
Title: Levothyroxine Treatment in Thyroid Benign Nodular Goiter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shyang-Rong, Shih, MD, National Taiwan University Hospital, Internal Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200612016M
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): under eltroxin
  Interventions: Drug: Levothyroxin treatment

INTERVENTIONS:
Drug: Levothyroxin treatment — Levothyroxin 100 micogram will be administered once daily 1 hour before meal of just after meal for 3 months, and the dose will be titrate to keep serum TSH level between 0.1~0.3 mU/L. It will be discontinued for 3 months. Then

SUMMARY:
We will study the effect of taking eltroxin at different time, i.e. fasting or postprandial periods. We will also study the effect of levothyroxin treatment in Chinese people

DETAILED DESCRIPTION:
OBJECTIVE - Current treatment of benign thyroid is oral levothyroxin by suppression of thyrotropin secretion and so that tumor growth. Although current consensus is taking thyroxin one hour before meal because the PH value of gastrointestinal tract will affect drug absorption, some patient suffered from epigastric discomfort when taking thyroxin with empty stomach, and wish to take it postprandial. However, there is no direct evidence showing if taking thyroxin at different time point significantly affects treatment outcome. Besides, the response to thyroxin therapy differs among people. The purposes of this study are to evaluate the clinical significance of different time points of thyroxine intake and to search factors relating to thyroxin response of benign thyroid tumors.

RESEARCH DESIGN AND METHODS - We will include patients who have benign thyroid tumors diagnosed with fine needle aspiration cytology and have normal thyroid function into our study. After informed consent, patients will be randomly assigned into two groups. Patients in the first group will take thyroxin one hour before breakfast until thyrotropin level stabilized between 0.5 and 1.0 mU/L for 3 months. Then thyroxin will be discontinued. Patients will restart thyroxin therapy three months later but after breakfast. Patients in another group will take thyroxin postprandial, discontinue thyroxin and then one hour before breakfast. Questionnaire interviews about diet and life style, blood samples and fine needle aspiration cytology samples will be obtained. Changes of thyroid nodules will be evaluated with thyroid echo.

STATISTIC ANALYSIS - Descriptive data will be described as means and SDs for continuous variables, and analysis of variance and Chi-square tests were used for assessing the significances. A p-value below 0.05 was considered significant.

Keywords: benign thyroid tumor, thyroxin, preprandial, postprandial.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 to 90 years old
2. Benign nodular goiter diagnosed with thyroid echo and fine-needle - aspiration cytology

Exclusion Criteria:

1. Age younger than 20 or older than 90 years old
2. Pregnancy
3. Allergy to eltroxin
4. Taking other drugs which will have drug interaction with eltroxin
5. patients with cardiovascular disease, hypertension, gastrointestinal disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The size of thyroid nodules | 3 months after levothyroxine treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shyang-Rong Shi, M.D., Principal Investigator — National Taiwan University Hospital, Yun-Lin Branch
Locations (1):
- National Taiwan University Hospital, Dou-Liou City, Yun-Lin County, Taiwan